CLINICAL TRIAL: NCT07037316
Title: Effect of Progressive Resistance Exercise With Lymphatic Taping Versus Progressive Resistance Exercise With Compression Bandages on Lymphedema in Pregnant Females
Brief Title: Effect of PRE With LT Versus PRE With Compression Bandages on Lymphedema in Pregnant Females
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1011
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- progressive resistance exercise with lymphatic taping (Experimental)
  Interventions: Diagnostic Test: progressive resistance exercise with lymphatic taping
- progressive resistance exercise with compression Bandage (Experimental)
  Interventions: Diagnostic Test: progressive resistance exercise with compression Bandage

INTERVENTIONS:
Diagnostic Test: progressive resistance exercise with lymphatic taping — Participants will receive a supervised, moderate-to-vigorous intensity resistance training program designed specifically for pregnant women, The resistance training will involve the use of light barbells (1-10 lbs) and weight plates (2.5-10 lbs), targeting all major muscle groups through 50-80 repetitions per muscle group over 3-5 minutes, with short rest intervals. Exercises will be performed at a self-rated intensity level considered moderate to vigorous, following the Borg scale for perceived exertion. The training program is based on the BodyPump format but modified to suit pregnancy-related safety considerations.
  Arms: progressive resistance exercise with lymphatic taping
Diagnostic Test: progressive resistance exercise with compression Bandage — Participants in will receive progressive resistance exercise same as Group B and also receive thecompression bandaging as the primary intervention for the management of lower-limb oedema during pregnancy. The compression bandage will be applied in a multi-layered manner, beginning from the base of the toes and extending proximally to below the knee, ensuring graded pressure with higher compression distally and gradually reducing proximally to support venous and lymphatic return. Prior to each application, participants will be asked to lie in a supine position with their legs elevated for 15-20 minutes to reduce pre-existing swelling.
  Arms: progressive resistance exercise with compression Bandage

SUMMARY:
This Study aims to compare the effectiveness of progressive resistance exercise (PRE) combined with lymphatic taping versus PRE combined with compression bandaging in managing lower limb lymphedema in pregnant women. Lymphedema during pregnancy is often caused by hormonal and mechanical changes that lead to fluid retention and swelling, significantly affecting mobility and quality of life. The study will involve 59 pregnant women diagnosed with lymphedema, divided into two groups.

DETAILED DESCRIPTION:
Both groups will follow a supervised PRE program, with one group receiving lymphatic kinesio taping and the other receiving compression bandaging as adjunct treatments. Outcomes will be assessed using the Visual Analog Scale (VAS) for pain, Borg scale for exertion, and Disability Rating Index for functional limitations. Data will be collected at baseline, week 4, and week 8.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females aged 18-40 years diagnosed with lymphedema.
* Nulliparous, primiparous, or multiparous pregnant females.
* resenting a sensation of heaviness, pain, swelling, and/or tingling in LL, with written authorization from their obstetrician.
* Ability to provide informed consent and comply with the treatment protocol.

Exclusion Criteria:

* pregnant women with some clinical instability, diagnosed with uncontrolled gestational hypertension, renal failure and deep vein thrombosis (DVT).
* Any Skin continuity, wound; dermatological, lymphatic, and cardiac diseases; infections; and voluminous and symptomatic varicose veins.
* High-risk pregnancy conditions such as placenta previa, preeclampsia, or any contraindications to exercise.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) | 6 Month
  A visual analog scale (VAS) score is determined by measuring the distance on a line, usually 10 centimeters long, where one end represents "no pain" and the other "worst pain
Disability Rating Index (DRI) | 6 Months
  The Disability Rating Index (DRI) is a tool used to assess the level of physical disability, with scores ranging from 0 to 100. A score of 0 represents normal function, while 100 indicates complete disability, according to ResearchGate. The Disability Rating Scale (DRS) is another measure, particularly for individuals with traumatic brain injuries, with scores ranging from 0 to 29, where higher scores indicate greater impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No